CLINICAL TRIAL: NCT05277428
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-design Clinical Study to Evaluate the Irritable Bowel Syndrome Symptoms Improving Effect and Safety of Lactobacillus Plantarum APsulloc 331261(GTB1)
Brief Title: Clinical Study to Evaluate the IBS Symptoms Improving Effect and Safety of GTB1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AP-AR-2020-1
Record Dates: First submitted 2022-02-21; First posted 2022-03-14 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Irritable Bowel Syndrome With Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus Plantarum APsulloc 331261(GTB1) (Experimental): Take GTB1 capsule once daily for 4 weeks
  Interventions: Dietary Supplement: GTB1
- Placebo (Placebo Comparator): Take placebo capsule once daily for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GTB1 — 2 capsule/day
  Arms: Lactobacillus Plantarum APsulloc 331261(GTB1)
Dietary Supplement: Placebo — 2 capsule/day
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of L. plantarum APsulloc 331261(GTB1TM) on improvement of IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 19 years old
* Diagnosed case of IBS using Rome IV criteria
* Who had type 6 or 7 stools according to the BSFS on at least 2 weeks ≥ 25%
* Who voluntarily agreed to participate in the study and signed an informed consent form

Exclusion Criteria:

* Who had been ingesting products containing probiotics or prebiotics in the 4 weeks preceding entry into the trial
* Who had antibiotic agents during the 4 weeks prior to study entry
* Women who is pregnant /breast-feeding, or who has childbearing potential and does not use available contraceptives
* Who is determined ineligible for study participation by investigators for any other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Changes in a global relief at 4 weeks | Global Relief after 4 weeks of ingestion
  Global relief of IBS is a dichotomous single item that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms?". The answer is YES or NO.
Changes in frequency and type of stools at 4 weeks from baseline | Baseline, and 4 weeks of ingestion
  Number of stools per day and type of stools assessed during 7 days before the visit. Type of stools assessed using the Bristol Stool Formation Scale.
Changes in severity and frequency of IBS-Intestinal discomfort symptoms at 4 weeks | Baseline, and 4 weeks of ingestion
  Intestinal discomfort symptoms are 3 symptoms that asks: abdominal pain, abdominal bloating, feeling of incomplete evacuation over the past 7 days.

SECONDARY OUTCOMES:
Changes in Quality of Life at 4 weeks from baseline | Baseline, 1, 2 and 4 weeks of ingestion
  Change of dissatisfaction with bowel habit and interfering with general life by Irritable Bowel Syndrome
Improvement or worsening of IBS global symptoms using Participants global impression of change scale and global improvement scale | Improvement/worsening assessed after 4 weeks of ingestion
  Improvement or worsening scale 1-7
Fecal microbiome | Baseline, 4 weeks of ingestion
  Changes in the fecal microbiome in participants with IBS-D due to use of GTB1

OTHER OUTCOMES:
Changes in a global relief | Global Relief after 1, 2 and 4 weeks of ingestion
  Global relief of IBS is a dichotomous single item that asks participants "Over the past week (7 days) have you had adequate relief of your IBS symptoms?". The answer is YES or NO.
Changes in frequency and type of stools | Baseline, 1, 2 and 4 weeks of ingestion and follow-up 2 weeks
  Number of stools per day and type of stools assessed during 7 days before the visit. Type of stools assessed using the Bristol Stool Formation Scale.
Changes in severity and frequency of IBS-Intestinal discomfort symptoms | Baseline, 1, 2 and 4 weeks of ingestion and follow-up 2 weeks
  Intestinal discomfort symptoms are 3 symptoms that asks: abdominal pain, abdominal bloating, feeling of incomplete evacuation over the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jonghwa Roh, PhD, Study Director — Amorepacific R&I center
Locations (1):
- Amorepacific, Yongin-si, Gyeonggi-do, South Korea